CLINICAL TRIAL: NCT06412627
Title: The Effect of Intervention About Dry Mouth and Thirst in Patients With Endotracheal Tube
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 231234
Record Dates: First submitted 2024-05-02; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Endotracheal Tube; Thirst; Dry Mouth
Keywords: dry mouth; thirst; endotracheal tube
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group received only usual care, while the Oral moisture checker (Mucus, Life Co., Ltd.), the Oral Health Assessment Tool, and the Bedside Oral Exam were used to assess oral mucosal moisture and oral health status before (day 0) and after 7 days.
- experimental group (Experimental): The experimental group had 4°C saline-soaked gauze applied to the oral cavity for 15 minutes at 06:00 AM and 06:00 PM daily for one week, while the Oral moisture checker (Mucus, Life Co., Ltd.), the Oral Health Assessment Tool, and the Bedside Oral Exam were used to assess oral mucosal moisture and oral health status before (day 0) and after 7 days.
  Interventions: Procedure: 4°C frozen normal saline gauze

INTERVENTIONS:
Procedure: 4°C frozen normal saline gauze — Soak two 4x4 gauze pads in 15 ml of normal saline, refrigerate at 4°C, and then apply in the oral cavity for 15 minutes before removal.
  Arms: experimental group

SUMMARY:
This is an experimental study aimed at exploring the effectiveness of using 4°C frozen gauze with normal saline for relieving dry mouth and thirst in patients with endotracheal tubes.

DETAILED DESCRIPTION:
Long-term placement of endotracheal tubes often causes discomfort, including lip ulcers, laryngeal pain, and dry oral mucosa, leading to frequent complaints of dry mouth and thirst among conscious patients. However, these symptoms are commonly overlooked in the nursing process, resulting in emotional distress and irritability in patients. Although healthcare providers recognize the issue of dry mouth and thirst in patients with endotracheal tubes, effective management is challenging due to concerns about treatment limitations, aspiration pneumonia, and the risk of coughing or vomiting. This experimental study aims to explore the effectiveness of using 4°C frozen gauze soaked in normal saline to relieve dry mouth and thirst in patients with endotracheal tubes.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal intubation.
* Aged 18 years or older.
* Patient or family members are willing to sign the consent form.

Exclusion Criteria:

* History of head and neck cancer.
* Oral mucosal damage, swelling, or bleeding that precludes placement of a moist gauze pad.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Oral moisture checking device | Change from baseline dry mouth at Day 3, and Day 7
  The oral moisture checking device was utilized to assess symptoms of dry mouth in participants.
  This study utilized an oral moisture checking device produced by Life Co., Ltd. of Japan, which measures the moisture content within the oral cavity using the principle of bioelectrical impedance analysis (BIA). The measurement method involves placing a specialized plastic sleeve over the tongue approximately one centimeter from the tip and applying a force of 200 grams. A measurement is obtained after about 2 seconds. A reading below 27.9 indicates dryness, a reading between 28 and 29.5 is considered borderline, and readings of 29.6 and above are normal. Both the sensitivity and specificity of this method are 0.8.

SECONDARY OUTCOMES:
Oral health assessment Tool | Change from baseline oral health status at Day 3, and Day 7
  The Oral health assessment Tool consists of 8 categories: lips, tongue, gum and tissues, saliva, natural teeth, dentures, oral cleanliness, and dental pain. The scoring is as follows: 0 points for "healthy," 1 point for "beginning changes in the mouth," and 2 points for "unhealthy." The maximum score is 16, with higher scores indicating poorer oral health.
Bedside oral examination scale | Change from baseline oral health function at Day 3, and Day 7
  The bedside oral examination scale comprises 8 categories: swallow, lips, tongue, mucous membranes, saliva, gingiva, teeth or dentures, and odor. Each category is scored as follows: 1 point for "severe dysfunction," 2 points for "moderate dysfunction," and 3 points for "normal." A total score of 24 indicates a normal oral health status, while a score of 8 indicates severe oral health dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan